CLINICAL TRIAL: NCT03189823
Title: Long-term Effect of Motor Cortex Stimulation in Patients Suffering From Chronic Neuropathic Pain
Acronym: MCSNL
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HenssenD
Record Dates: First submitted 2017-06-07; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Pain, Intractable; Central Pain Syndrome; Facial Pain
MeSH Terms: conditions — Pain, Intractable; Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Specify, model 3998, Medtronic Inc., Minneapolis, MN, USA — In MCS, an electrode is placed perpendicular to the central sulcus in the epidural space (Specify, model 3998, Medtronic Inc., Minneapolis, MN, USA) in order to obtain pain relief.
  Other Names: Motor cortex stimulation

SUMMARY:
In order to create insights in the effects of Motor cortex stimulation (MCS) on intractable pain, an open observational study was started in 2003. The aim of this research is to:

1. to determine the clinical effectivity of MCS on pain intensity after 1 month, 1 year and 3 years of stimulation
2. to determine the clinical effectivity of MCS on QoL and daity medication intake after 3 years of MCS

DETAILED DESCRIPTION:
2.1 Study protocol In 2003, an observational study protocol was set up in the university medical centers of Nijmegen and Groningen, the Netherlands, in order to study the effects of MCS in patients that suffered from chronic neuropathic pain. Patients were included between 2005 and 2013 when they suffered from chronic intractable pain and reported high levels of pain (VAS > 5, measured three times daily during four days) and when the chronic neuropathic pain had showed to be intractable. Furthermore, on radiographic imaging techniques performed less than three years before inclusion for the implantation of MCS should show a possible conflict that might contribute to the pain. A multidisciplinary approach by the anesthesiologist-pain specialists, neurosurgeons, and clinical psychologists was chosen for the selection of patients. Patients with severe, current psychological problems (e.g., depression, high anxiety) or substance-abuse were excluded. Other exclusion criteria were the use of therapeutic anticoagulants, cognitive and/or psychiatric disorders in the medical history, nociceptive pain, an expected life expectancy less than 3 years due to other diseases (e.g., cancer), contra- indications for general anesthesia (e.g., severe cardio-pulmonal diseases), convulsive disorders and the presence of other neuromodulation systems. All patients underwent preoperative somatosensory-evoked potential (SSEP) measurement to determine the integrity of the somatosensory system in order to facilitate intra-operative neurophysiological monitoring. A MRI-scan was used to determine any anatomical contra-indications (brain atrophy, pathological structures) for the operative procedure. All patients presented in this study had a follow up of three years.

2.2 Surgical technique The pre-operative fMRI was fused with the neuronavigation MRI. For this purpose, cortex surface rendering technique was performed using the Stealthviz software (Medtronic Inc., Minneapolis, MN, USA) to visualize the cortical areas and determine the central sulcus and the motor cortex, which then was marked on the skin by using neuronavigation. All patients were operated under general anesthesia without muscle relaxation. A small craniotomy (approximately 4 × 4 cm) was carried out over the central sulcus. An electrode was placed perpendicular to the central sulcus in the epidural space (Specify, model 3998, Medtronic Inc., Minneapolis, MN, USA). A phase-reversal somatosensory-evoked potential was used to confirm the position of the central sulcus, thereafter cortical stimulation was performed to map functional motor areas. Following identification of the optimal target, the electrode was sutured to the dura mater. After placement of the electrode, the electrode was tunneled subcutaneously and connected with an internalized pulse generator (IPG) (Medtronic Versitrel and later Prime Advanced) that was implanted in the subclavian space or in a subcutaneous abdominal pocket.

2.3 Data-analysis An independent researcher, who was blinded to the stimulation conditions, investigated the patient records in this observational study. Only patients who were treated in accordance to the aforementioned treatment protocol and with a minimal follow-up of three years in whom the effect of MCS, occurrence of complications, daily intake of medication and change in quality of life was complete, were analyzed.

2.4 Ethical statement and registration of clinical trial This observational study was performed under the approval of the medical ethical committee of the region Arnhem-Nijmegen. All patients, after extensive pre-operative information, gave written informed consent due to the experimental nature of this treatment at that time. This clinical trial was not registered in 2003 due to the fact that, in The Netherlands, MCS was not an experimental method at that moment. The authors confirm that all ongoing and related trials for this intervention are registered

2.5 Assessment Pain is a complex, subjective and multidimensional phenomenon that is difficult to measure by unidimensional pain scores only. Apart from the visual analog scale (VAS), the intake of pain medication is thought to be a valid tool of measuring pain relief. Adding analgesic drug intake as an outcome parameter could provide a more realistic assessment of long-term benefits of MCS. Four outcome variables were examined: 1) the amount of pain relief, measured by the mean difference between VAS score pre-operatively and the VAS score during the follow-up (1 month, 6 months, 1 year, and 3 years after implantation of the MCS electrodes); 2) the change in the drug regimen of all patients per day; 3) adverse events (infection, bleeding, hardware removal, temporary seizures, and battery dysfunction); and 4) the correlation between stimulation parameters and the pain relief per patient. Pain relief was divided into three categories. A good pain relief, level 1, was defined as a VAS reduction of 70-100%. Reduction of pain according to a VAS scores change between 40% and 69% was defined as satisfactory (level 2), while a minimal pain relief was defined as a reduction of ≤ 40% on the VAS scores. An effective pain relief was defined as ≥ 40% reduction of pain (levels 1 and 2). The use of medication was monitored using the electronic patient record during follow-up. The medication quantification scale (MQS) was used in order to quantify medication use and was calculated for each drug by multiplying the dosage levels by their respective detriment weight. The dosage levels (0-6) were based on the recommended daily dosage range as described by Masters Steedman et al. These scores are summed to provide a quantitative index of total drug intake suitable for statistical analysis. The occurrence of complications was documented as well. Apart from biological complications (eg. bleeding, infection), the removal of the hardware due to a minimal effect was evaluated as well. To determine whether there was a correlation between the used stimulation parameters and the pain relief, the used stimulation parameters (intensities [V], pulse widths [µs], and frequencies [Hz]) were reviewed. Interference of pain with quality of life (QoL) was measured before and after (> 1 year) MCS with use of the Quality of Life Index (QLI), based on the Dutch version of the McGill pain questionnaire (MPQ-DLV).

2.6 Statistical analysis IBM SPSS Statistics version 22 was used for statistical analyses of the retrieved data (IBM Corp. Released 2013. IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY: IBM Corp.). To analyze the differences in pain relief and MQS scores and QoL-indices per subgroup, the Mann-Whitney U test was used. In order to correlate the applied stimulation parameters, the Spearman rank correlation coefficient was conducted. Values are represented as mean ± standard deviation (minimum- maximum). Alterations in MQS scores and QoL-indices before and after MCS were calculated with use of the Wilcoxon signed-rank test. Statistical tests were two sided and with a significance level of P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Patients were included between 2005 and 2013 when they suffered from chronic intractable pain and reported high levels of pain (VAS > 5, measured three times daily during four days) and when the chronic neuropathic pain had showed to be intractable. Furthermore, on radiographic imaging techniques performed less than three years before inclusion for the implantation of MCS should show a possible conflict that might contribute to the pain. A multidisciplinary approach by the anesthesiologist-pain specialists, neurosurgeons, and clinical psychologists was chosen for the selection of patients.

Exclusion Criteria:

Patients with severe, current psychological problems (e.g., depression, high anxiety) or substance-abuse were excluded. Other exclusion criteria were the use of therapeutic anticoagulants, cognitive and/or psychiatric disorders in the medical history, nociceptive pain, an expected life expectancy less than 3 years due to other diseases (e.g., cancer), contra- indications for general anesthesia (e.g., severe cardio-pulmonal diseases), convulsive disorders and the presence of other neuromodulation systems.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Dutch patients that suffered from chronic, intractable neuropathic pain
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | 1month, 6months, 1 year and 3 years postoperative
  According to VAS scores

SECONDARY OUTCOMES:
Changes in quality of life | 3 years postoperative
  Interference of pain with quality of life (QoL) was measured before and after (> 1 year) MCS with use of the Quality of Life Index (QLI), based on the Dutch version of the McGill pain questionnaire (MPQ-DLV)
Changes in daily medication intake | 3 years postoperative
  The use of medication was monitored using the (electronic) patient record before MCS and during follow-up. The medication quantification scale (MQS) was used in order to quantify medication use and was calculated for each drug by multiplying the dosage levels by their respective detriment weight(21). The dosage levels (0-6) were based on the recommended daily dosage range as described by Masters Steedman et al.(22). These scores are summed to provide a quantitative index of total drug intake suitable for statistical analysis.

OTHER OUTCOMES:
Occurence of complications | during 3 years postoperative
  The occurrence of complications was documented as well. Apart from biological complications (eg. bleeding, infection), the removal of the hardware due to a minimal effect was evaluated as well using the (electronic) patient record

IPD SHARING:
Plan to Share IPD: Yes
An anominized excel file, compatible with SPSS will be attached to the submitted manuscript

REFERENCES:
- See also: Protocol in Dutch — http://www.imsn.nl/neuromod/MCS060104.pdf